CLINICAL TRIAL: NCT07315828
Title: A Prospective Study on the Accuracy of Indocyanine Green Fluorescence Imaging for the Visualization of Residual Lesions in the Tumor Cavity During Surgery for Giant Cell Tumor of Bone
Brief Title: Accuracy of Indocyanine Green (ICG) Fluorescence Imaging in Giant Cell Tumor of Bone Surgery
Acronym: ICG-GCTB
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other)
Responsible Party: Principal Investigator, Qingcheng Yang, Chief Orthopaedic Surgeon & Director, Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025-146; 2025-146 (Other: Ethics Committee of Shanghai Sixth People's Hospital)
Record Dates: First submitted 2025-12-20; First posted 2026-01-02 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2026-01

CONDITIONS: Giant Cell Tumor of Bone
Keywords: Indocyanine Green; Fluorescence Imaging; Near-Infrared Imaging; Giant Cell Tumor of Bone
MeSH Terms: conditions — Giant Cell Tumor of Bone | interventions — Indocyanine Green

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-center, single-arm study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICG Fluorescence Imaging Group (Experimental): All enrolled participants receive ICG fluorescence-guided surgery. Following standard tumor curettage, the bone cavity is systematically explored using a near-infrared fluorescence imaging system. The intervention consists of detecting residual fluorescence signals, obtaining verification samples for blinded pathological assessment, and performing supplementary curettage of confirmed suspicious lesions to achieve potentially cleaner surgical margins.
  Interventions: Drug: Indocyanine Green

INTERVENTIONS:
Drug: Indocyanine Green — Participants receive an intravenous injection of Indocyanine Green (ICG) at a dose of 0.25-0.5 mg/kg, 1-6 hours prior to surgery. Intraoperatively, a near-infrared fluorescence imaging system is used to guide the exploration of the bone cavity. The intervention involves a "verify first, treat later" protocol: it includes diagnostic verification sampling of fluorescence-positive areas and, crucially, therapeutic supplementary curettage of residual fluorescent lesions that were missed during standard white-light surgery.
  Other Names: ICG

SUMMARY:
This study evaluates the diagnostic accuracy of Indocyanine Green (ICG) fluorescence imaging in visualizing residual lesions of Giant Cell Tumor of Bone (GCTB) in the tumor cavity during surgery. Patients diagnosed with GCTB will receive an intravenous injection of ICG prior to the operation to label tumor tissues. During the procedure, surgeons will use a near-infrared fluorescence imaging system to visualize the tumor cavity and identify potential residual lesions after standard curettage. The study aims to determine the sensitivity, specificity, positive predictive value, and negative predictive value of ICG fluorescence imaging by comparing the intraoperative fluorescence findings with the final pathological results of the validation samples.

DETAILED DESCRIPTION:
Giant Cell Tumor of Bone (GCTB) poses a significant surgical challenge due to the difficulty in detecting microscopic residual tumor tissues in the bone cavity, which contributes to a high local recurrence rate. This prospective, single-center, single-arm study aims to evaluate the accuracy of Indocyanine Green (ICG) fluorescence imaging in visualizing GCTB lesions during surgery. Eligible patients will receive an intravenous injection of ICG (0.25-0.5 mg/kg) 1-6 hours before surgery. Following standard tumor curettage under white light, the bone cavity will be systematically explored using a near-infrared fluorescence imaging system to visualize potential residual tumor tissues. The surgeon will obtain validation samples from fluorescence-positive areas, fluorescence-negative background tissues, and post-treatment beds for blinded pathological assessment. The study will quantify the diagnostic performance of ICG imaging by calculating sensitivity, specificity, positive predictive value, and negative predictive value based on the pathological gold standard, alongside secondary analyses of tumor-to-background ratios and microscopic tumor boundary concordance.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Giant Cell Tumor of Bone(GCTB), via preoperative biopsy or typical imaging (MRI), and scheduled for surgical resection.
* Capable of understanding the study and voluntarily signing the written informed consent form.

Exclusion Criteria:

* Known severe history of allergy to Indocyanine Green (ICG) or iodine.
* Severe liver dysfunction.
* Women who are pregnant or lactating.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy of ICG Fluorescence Imaging (Sensitivity, Specificity, PPV, NPV) | From the time of surgery until the final pathology report is available, assessed up to 1 week post-operatively.
  The diagnostic performance of ICG fluorescence imaging in detecting GCTB lesions will be evaluated by comparing the intraoperative fluorescence status (Positive/Negative) with the final histopathological diagnosis (Tumor/Non-tumor) of the resected specimens. The unit of analysis is the individual specimen. The following metrics will be calculated: Sensitivity, Specificity, Positive Predictive Value (PPV), and Negative Predictive Value (NPV).

SECONDARY OUTCOMES:
Tumor-to-Background Ratio (TBR) | Intraoperative
  TBR is a quantitative measure of fluorescence intensity. It will be calculated by dividing the mean fluorescence intensity of the tumor region by the mean fluorescence intensity of the adjacent normal background tissue using image analysis software.
Incidence of ICG-Related Adverse Events | From the time of ICG injection through 24 hours post-surgery
  The number of participants experiencing adverse events related to ICG administration (e.g., allergic reactions, anaphylactic shock) will be monitored and recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Sixth People's Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nicoli F, Saleh DB, Baljer B, Chan CD, Beckingsale T, Ghosh KM, Ragbir M, Rankin KS. Intraoperative Near-infrared Fluorescence (NIR) Imaging With Indocyanine Green (ICG) Can Identify Bone and Soft Tissue Sarcomas Which May Provide Guidance for Oncological Resection. Ann Surg. 2021 Feb 1;273(2):e63-e68. doi: 10.1097/SLA.0000000000003857. PMID 32224746
- [Result] Wang H, Ji T, Qu H, Yan T, Li D, Yang R, Tang X, Guo W. Indocyanine green fluorescence imaging may detect tumour residuals during surgery for bone and soft-tissue tumours. Bone Joint J. 2023 May 1;105-B(5):551-558. doi: 10.1302/0301-620X.105B5.BJJ-2022-0803.R1. PMID 37121591
- [Result] Huang H, He S, Wei R, Zhu X, Deng Z, Wang Y, Guo L, Lei J, Cai L, Xie Y. Near-infrared (NIR) imaging with indocyanine green (ICG) may assist in intraoperative decision making and improving surgical margin in bone and soft tissue tumor surgery. J Surg Oncol. 2023 Sep;128(4):612-627. doi: 10.1002/jso.27306. Epub 2023 May 13. PMID 37178368
- [Result] Vinegoni C, Botnaru I, Aikawa E, Calfon MA, Iwamoto Y, Folco EJ, Ntziachristos V, Weissleder R, Libby P, Jaffer FA. Indocyanine green enables near-infrared fluorescence imaging of lipid-rich, inflamed atherosclerotic plaques. Sci Transl Med. 2011 May 25;3(84):84ra45. doi: 10.1126/scitranslmed.3001577. PMID 21613624
- [Result] Newton AD, Predina JD, Shin MH, Frenzel-Sulyok LG, Vollmer CM, Drebin JA, Singhal S, Lee MK 4th. Intraoperative Near-infrared Imaging Can Identify Neoplasms and Aid in Real-time Margin Assessment During Pancreatic Resection. Ann Surg. 2019 Jul;270(1):12-20. doi: 10.1097/SLA.0000000000003201. PMID 31188797
- [Result] Dip F, Boni L, Bouvet M, Carus T, Diana M, Falco J, Gurtner GC, Ishizawa T, Kokudo N, Lo Menzo E, Low PS, Masia J, Muehrcke D, Papay FA, Pulitano C, Schneider-Koraith S, Sherwinter D, Spinoglio G, Stassen L, Urano Y, Vahrmeijer A, Vibert E, Warram J, Wexner SD, White K, Rosenthal RJ. Consensus Conference Statement on the General Use of Near-infrared Fluorescence Imaging and Indocyanine Green Guided Surgery: Results of a Modified Delphi Study. Ann Surg. 2022 Apr 1;275(4):685-691. doi: 10.1097/SLA.0000000000004412. PMID 33214476
- [Result] Machak GN, Snetkov AI. The impact of curettage technique on local control in giant cell tumour of bone. Int Orthop. 2021 Mar;45(3):779-789. doi: 10.1007/s00264-020-04860-y. Epub 2020 Oct 22. PMID 33094400
- [Result] Aoude A, Nikomarov D, Perera JR, Ibe IK, Griffin AM, Tsoi KM, Ferguson PC, Wunder JS. Giant cell tumour of bone. Bone Joint J. 2023 May 1;105-B(5):559-567. doi: 10.1302/0301-620X.105B5.BJJ-2022-1231.R1. PMID 37121582
- [Result] Basu Mallick A, Chawla SP. Giant Cell Tumor of Bone: An Update. Curr Oncol Rep. 2021 Mar 22;23(5):51. doi: 10.1007/s11912-021-01047-5. PMID 33754215
- [Result] Werner M. Giant cell tumour of bone: morphological, biological and histogenetical aspects. Int Orthop. 2006 Dec;30(6):484-9. doi: 10.1007/s00264-006-0215-7. Epub 2006 Sep 30. PMID 17013643